CLINICAL TRIAL: NCT02623036
Title: The Use of Ambulatory Blood Pressure Monitors to Assess Angiotensin Converting Enzyme Inhibitors in Resistant Hypertension
Brief Title: The Use of Ambulatory Blood Pressure Monitors to Assess Angiotensin Converting Enzyme Inhibitors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Memorial Health University Medical Center (Other)
Responsible Party: Principal Investigator, John Bucheit, Pharm.D.,BCACP, CDE, Principal Investigator, Memorial Health University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHUMC 2015.10.01
Record Dates: First submitted 2015-11-19; First posted 2015-12-07 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Hypertension, Resistant to Conventional Therapy
Keywords: chronotherapy; angiotensin converting enzyme inhibitors; ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy | interventions — Enalaprilat; Lisinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enalapril arm (Active Comparator): Patients randomized to this group will receive equivalent dose enalapril to their current ACEI therapy and change the administration time to bedtime.
  Interventions: Drug: Equivalent dose enalapril
- Lisinopril arm (Active Comparator): Patients randomized to this group will receive equivalent dose lisinopril to their current ACEI therapy and change the administration time to bedtime.
  Interventions: Drug: Equivalent dose lisinopril

INTERVENTIONS:
Drug: Equivalent dose enalapril — Chronotherapy with enalapril.
  Other Names: Vasotec
  Arms: Enalapril arm
Drug: Equivalent dose lisinopril — Chronotherapy with lisinopril
  Other Names: Prinivil
  Arms: Lisinopril arm

SUMMARY:
The purpose of this study is to use ambulatory blood pressure monitors to investigate whether enalapril is superior to lisinopril in managing nocturnal hypertension in patients with resistant hypertension currently treated with daytime angiotensin converting enzyme inhibitors.

DETAILED DESCRIPTION:
Resistant hypertension is defined as blood pressure > 140/90 mm Hg while adherent to three or more antihypertensive medications or < 140/90 mm Hg treated with four or more antihypertensives. Patients with resistant hypertension may be at risk for elevated nighttime blood pressure >120/70 mm Hg and "non-dipping" (night/day blood pressure > 0.9). A higher rate of cardiovascular events occur during the "morning surge" partially attributed elevated nighttime blood pressure due to increased renin angiotensin aldosterone system (RAAS) activity. Angiotensin converting enzyme inhibitors (ACEIs) suppress RAAS activity

This prospective randomized parallel-group pilot study will occur at Memorial Family Medicine. Eligible patients will undergo three study visits over a 5-8 week span. After providing written informed consent, patients will complete an initial screening visit assessing 25 hour blood pressure using ambulatory blood pressure monitors. Patients will continue the study if they are found to have a nighttime blood pressure >120/70 mm Hg. Patients continuing the study will be randomly assigned to equivalent dose lisinopril or enalapril treatment arms and their administration time will be changed to "bedtime." At the final visit, patients will complete a final ambulatory blood pressure analysis to reassess nighttime blood pressure and dipping status.

It's expected that patients with enalapril treatment will have superior nighttime blood pressure reduction compared to the lisinopril treatment group. If the expected outcome occurs, more patients in the enalapril group will meet their nighttime blood pressure goal (<120/70 mm Hg) and exhibit a "dipping pattern." Current evidence suggests that patients with normal nighttime blood pressure and dipping pattern are at a lower risk for cardiovascular morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinic blood pressure > 140/90 mm Hg on 3 antihypertensives or clinic blood pressure < 140/90 mm Hg on 4 antihypertensives
* Currently treated with an angiotensin converting enzyme inhibitor

Exclusion Criteria:

* Chronic kidney disease (CKD) stage 4 or worse
* Pheochromocytoma
* Unstable cardiovascular disease Stroke, Transient Ischemic Attack, Unstable Angina, or Myocardial infarction in the last 30 days
* Hyperaldosteronism
* Current pregnancy
* Shift worker at night
* Presenting blood pressure > 180/110 mm Hg

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline nighttime blood pressure | Baseline and 4-6 weeks
  Average blood pressure between 0000-0600.

SECONDARY OUTCOMES:
Change from baseline night to day blood pressure ratio (dipping status) | Baseline and 4-6 weeks
  Nighttime blood pressure (average 0000-0600)/Daytime blood pressure 0900-2100. This outcomes evaluates patients' circadian blood pressure pattern. A normal circadian blood pressure pattern shows a 10% decrease in both systolic and diastolic blood pressure at night. This will help measure the impact of chronotherapy between the 2 study agents.
Change from baseline 24 Hour Blood Pressure | Baseline and 4-6 weeks
  Average blood pressure over 24 hours (0000-2359)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Bucheit, Pharm D, Principal Investigator — Memorial Health University Medical Center
Locations (1):
- Memorial Family Medicine Center, Savannah, Georgia, United States

REFERENCES:
- [Background] Calhoun DA, Jones D, Textor S, Goff DC, Murphy TP, Toto RD, White A, Cushman WC, White W, Sica D, Ferdinand K, Giles TD, Falkner B, Carey RM; American Heart Association Professional Education Committee. Resistant hypertension: diagnosis, evaluation, and treatment: a scientific statement from the American Heart Association Professional Education Committee of the Council for High Blood Pressure Research. Circulation. 2008 Jun 24;117(25):e510-26. doi: 10.1161/CIRCULATIONAHA.108.189141. PMID 18574054
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- [Result] Weisser K, Schloos J, Lehmann K, Dusing R, Vetter H, Mutschler E. Pharmacokinetics and converting enzyme inhibition after morning and evening administration of oral enalapril to healthy subjects. Eur J Clin Pharmacol. 1991;40(1):95-9. doi: 10.1007/BF00315146. PMID 1647954